CLINICAL TRIAL: NCT05650333
Title: AN INTERVENTIONAL PK, PD, PHASE 1, OPEN-LABEL STUDY TO INVESTIGATE PK AND PD OF MULTIPLE-DOSE RITLECITINIB IN CHILDREN 6 TO LESS THAN 12 YEARS OF AGE WITH SEVERE ALOPECIA AREATA
Brief Title: A Study to Learn About the Study Medicine (Called Ritlecitinib) For the Potential Treatment of Severe Alopecia Areata (AA) In Children 6 To Less Than 12 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B7981031
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-06

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ritlecitinib 20 mg (Experimental): Participants will receive Ritlecitinib 20 mg by mouth once daily (QD).
  Interventions: Drug: Ritlecitinib 20 mg

INTERVENTIONS:
Drug: Ritlecitinib 20 mg — orally administered, Ritlecitinib 20 mg once daily (QD)

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics (how the medicine is changed and eliminated from your body after you take it) and pharmacodynamics (effects of the medicine in the body) of the study medicine (called Ritlecitinib) in children of 6 to <12 years of age with Alopecia Areata, a condition of scalp hair loss. 12 children with alopecia areata will be participating in this study. All participants will receive study medicine with a dose of 20 milligram (mg) orally once daily for 7 days. 5 blood samples will be collected on day 7 for pharmacokinetic evaluation and 2 blood samples each at screening and on Day 7 will be collected for pharmacodynamic evaluation. Participants will take part in the study for about 10 weeks.

DETAILED DESCRIPTION:
This is an interventional, Pharmacokinetic (PK), Pharmacodynamic (PD), phase 1, open label study in children 6 to less than 12 years of age with ≥50% scalp hair loss due to severe alopecia areata. The purpose of the study is to collect data to support dose selection for subsequent studies in the same population.

Participants will be screened and, if all eligibility criteria are met, will receive the first dose of Investigational product within 28 days after the screening visit.

Participants will receive 20 mg ritlecitinib in one dose, daily, for 7 consecutive days. Blood samples for pharmacodynamic evaluation will be collected on screening and Day 7. Blood samples for pharmacokinetic evaluation will be collected on Day 7 at: 0 hr (pre-dose), 0.5 hr, 1 hr, 3 hrs, and 8 hrs after dosing.

At least 12 evaluable participants with respect to the primary endpoint will be enrolled in the study.

Participants and their parents/legal guardians will be required to visit the study site 3 times during the study (Screening, Day 1 and Day 7) A safety follow-up visit will be conducted by phone, 28 to 35 days after the last dose of ritlecitinib.

ELIGIBILITY:
Key Inclusion criteria:

1. Participants who are 6 to less than12 years old at the baseline visit.
2. A diagnosis of severe AA, including AT and AU, with ≥50% scalp hair loss due to AA (ie, a SALT score of ≥50) at both the Screening and Baseline visits, without evidence of terminal hair regrowth within the previous 12 months.

Key Exclusion Criteria:

1. A known congenital cause of AA, other systemic diseases that may cause hair loss (eg, lupus erythematosus, thyroiditis, systemic sclerosis, lichen planus, etc) or other etiology of hair loss (eg, telogen effluvium, androgenetic alopecia, etc).
2. Any present malignancies or history of malignancies, history of any lymphoproliferative disorder
3. History (one or more episodes) of CMV, varicella, herpes zoster (shingles) or disseminated herpes simplex.
4. Other medical or psychiatric condition (including recent [within the past year] or active suicidal ideation/behavior) that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
5. Not up to date with all age appropriate vaccines (including 2-dose vaccination for varicella) or vaccination with attenuated live vaccine within 6 weeks of first dose of study medicine.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (9):
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Pediatric Skin Research,LLC, Coral Gables, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - UNMH, Albuquerque, New Mexico
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Northwest Dermatology Institute, Portland, Oregon
  - Texas Dermatology and Laser Specialists, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Gonzalez ME, Browning J, Smith S, Plotka A, Zhu JD, Parvatini S, Huh Y, Wolk R. A Phase 1, Open-Label Study of the Pharmacokinetics of Ritlecitinib in Children Aged 6-12 Years With Alopecia Areata. Pediatr Dermatol. 2025 Jul-Aug;42(4):742-746. doi: 10.1111/pde.15895. Epub 2025 Feb 9. PMID 39924925
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981031

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 15 participants, 6 to less than 12 years of age with greater than or equal to (>=) 50% scalp hair loss due to alopecia areata, were enrolled. Study started from 02 March 2023 and completed on 11 August 2023.
Groups:
- Ritlecitinib 20 mg: Participants received Ritlecitinib 20 milligram (mg) orally once daily (QD), for 7 consecutive days. Participants were followed up to 35 days after the last dose.
Period: Treatment Period (7 Days)
Arm/Group | Ritlecitinib 20 mg
Started | 15
Completed | 14
Not Completed | 1
Not completed — Adverse Event | 1
Period: Follow-up (35 Days After Last Dose)
Arm/Group | Ritlecitinib 20 mg
Started | 15 (All enrolled participants were followed-up.)
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in the study and were assigned to study intervention.
Groups:
- Ritlecitinib 20 mg: Participants received Ritlecitinib 20 mg orally QD, for 7 consecutive days. Participants were followed up to 35 days after the last dose.
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.5 (1.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Profile Over the Dosing Interval of 24 Hours, at Steady State (AUC24ss/AUCtau) of Ritlecitinib on Day 7
Description: Linear-log trapezoidal method was used for evaluation. For the calculation of AUCtau, pre-dose concentration of Day 7 was used as an estimate for the concentration of 24 hours post-dose on Day 7.
Time Frame: Day 7: 0 (pre-dose), 0.5, 1, 3, 8 and 24 hours [pre-dose concentration was used as an estimate for the concentration of 24 hours post dose]
Population: Pharmacokinetic (PK) parameter analysis population: treated participants who had at least 1 of the PK parameters of primary interest. All participants with evaluable PK were included in the analysis. Two participants weren't included in analysis as they didn't have evaluable PK data (1 discontinued study intervention on Day 3 and the other had the important protocol deviation, PK samples not collected on Day 7). "Number of Participants Analyzed": participants evaluable for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hours per milliliter (ng*hr/mL)
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 13
Nanogram*hours per milliliter (ng*hr/mL) | 437.5 (30) [lower limit 30]

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ritlecitinib
Time Frame: 0 (pre-dose), 0.5, 1, 3 and 8 hours post-dose on Day 7
Population: PK parameter analysis population: treated participants who had at least 1 of the PK parameters of primary interest. All participants with evaluable PK were included in the analysis. Two participants weren't included in analysis as they didn't have evaluable PK data (1 discontinued study intervention on Day 3 and the other had the important protocol deviation, PK samples not collected on Day 7). "Number of Participants Analyzed": participants evaluable for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 13
Nanogram per milliliter (ng/mL) | 208.7 (38) [lower limit 38]

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Ritlecitinib
Time Frame: 0 (pre-dose), 0.5, 1, 3 and 8 hours post-dose on Day 7
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 13
Hours | 0.500 (0.450) [0.450 to 1.00]

4. Secondary Outcome: Apparent Oral Clearance (CL/F) of Ritlecitinib
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological process. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: 0 (pre-dose), 0.5, 1, 3 and 8 hours post-dose on Day 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 13
Liter per hour (L/hr) | 45.70 (30) [lower limit 30]

5. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Ritlecitinib
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/F is influenced by the fraction absorbed.
Time Frame: 0 (pre-dose), 0.5, 1, 3 and 8 hours post-dose on Day 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 8
Liter | 74.92 (23) [lower limit 23]

6. Secondary Outcome: Elimination Half-Life (t1/2) of Ritlecitinib
Description: Elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by one half at the elimination phase.
Time Frame: 0 (pre-dose), 0.5, 1, 3 and 8 hours post-dose on Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 8
Hours | 1.191 (0.10776) [lower limit 0.10776]

7. Secondary Outcome: Change From Baseline in Interferon Gamma Induced Protein 10 (IP-10) on Day 7
Time Frame: Baseline and Day 7
Population: The pharmacodynamic (PD) parameter analysis population included all participants treated who had at least 1 of the PD parameters of primary interest. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Median (Full Range); unit: Picogram per milliliter (pg/mL)
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 15
Picogram per milliliter (pg/mL)
  Baseline | 121.0 [74.7 to 888.0]
  Change at Day 7: number analyzed (Participants) | 12
  Change at Day 7 | -9.9 [-555.0 to 104.0]

8. Secondary Outcome: Change From Baseline in T Lymphocytes on Day 7
Description: T lymphocytes included CD3 cells, CD4 T helper lymphocytes and CD8 T cytotoxic lymphocytes.
Time Frame: Baseline and Day 7
Population: The PD parameter analysis population included all participants treated who had at least 1 of the PD parameters of primary interest. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Median (Full Range); unit: 10^9 cells per liter
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 15
10^9 cells per liter
  CD3 cells: Baseline | 1.8 [0.8 to 3.4]
  CD3 cells: Change at Day 7: number analyzed (Participants) | 12
  CD3 cells: Change at Day 7 | -0.0 [-1.3 to 2.0]
  CD4 T helper lymphocytes: Baseline | 1.0 [0.6 to 1.6]
  CD4 T helper lymphocytes: Change at Day 7: number analyzed (Participants) | 12
  CD4 T helper lymphocytes: Change at Day 7 | -0.1 [-0.6 to 1.1]
  CD8 T cytotoxic lymphocytes: Baseline | 0.6 [0.2 to 1.5]
  CD8 T cytotoxic lymphocytes: Change at Day 7: number analyzed (Participants) | 12
  CD8 T cytotoxic lymphocytes: Change at Day 7 | 0.0 [-0.6 to 0.8]

9. Secondary Outcome: Change From Baseline in B Lymphocytes on Day 7
Description: B lymphocytes included CD19 cells.
Time Frame: Baseline and Day 7
Population: as for outcome 8
Measure: Median (Full Range); unit: 10^6 cells per liter
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 15
10^6 cells per liter
  Baseline | 439.0 [191.0 to 881.0]
  Change at Day 7: number analyzed (Participants) | 12
  Change at Day 7 | -19.0 [-116.0 to 766.0]

10. Secondary Outcome: Change From Baseline in Natural Killer (NK) Cells on Day 7
Time Frame: Baseline and Day 7
Population: as for outcome 8
Measure: Median (Full Range); unit: 10^6 cells per liter
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 15
10^6 cells per liter
  Baseline | 254.0 [85.0 to 729.0]
  Change at Day 7: number analyzed (Participants) | 12
  Change at Day 7 | -25.5 [-318.0 to 627.0]

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Treatment-emergent were events between first dose to 35 days after last dose, that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Day 1 of dosing up to 35 days after the last dose (maximum up to Day 42)
Population: Safety analysis set included all participants assigned to study intervention and who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 15
Participants | 3

12. Secondary Outcome: Number of Participants With Treatment Related AEs
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Relatedness was judged by investigator.
Time Frame: Day 1 of dosing up to 35 days after the last dose (maximum up to Day 42)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 15
Participants | 1

13. Secondary Outcome: Number of Participants With Serious AEs (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Day 1 of dosing up to 35 days after the last dose (maximum up to Day 42)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 15
Participants | 0

14. Secondary Outcome: Number of Participants With AEs Leading to Treatment Discontinuation
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Day 1 up to Day 7
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 15
Participants | 1

15. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital signs evaluation included blood pressure and heart rate measurements. Clinical significance of any vital sign abnormality was judged by investigator.
Time Frame: Day 1 up to Day 7
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 15
Participants | 0

16. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Values
Description: Clinical laboratory parameters included haematology: haemoglobin, haematocrit, red blood cells count, platelet count, white blood cells count, total absolute: neutrophils, eosinophils, monocytes, basophils, lymphocytes; chemistry: urea and creatinine estimated creatinine clearance, glucose (fasting), sodium, potassium, chloride, aspartate aminotransferase (AT), alanine AT, total bilirubin, alkaline phosphatase, albumin, total protein; urinalysis: local dipstick: pH, qualitative: glucose, protein, albuminuria, blood, ketones, nitrites, leukocyte esterase and others. Clinical significance of any laboratory abnormality was judged by investigator.
Time Frame: Day 1 up to Day 7
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 15
Participants | 0

17. Secondary Outcome: Number of Participants as Per Score for Pediatric Taste Assessment Questionnaire
Description: The pediatric taste questionnaire included 3 questions regarding: 1) Overall Taste (likeability in tase), 2) Overall Mouthfeel (how the medicine felt) and 3) Overall Volume of Medicine (likeability of the amount of medicine). Each question ranged from 1 (most favorable) to 5 (least favorable), higher scores indicates less liking to medicine. Ritlecitinib was provided as capsules; for administration, the capsules were dissolved in water and the contents of the capsule in water were taken according to the dosing administration instructions.
Time Frame: Day 1 and 7
Population: Safety analysis set included all participants assigned to study intervention and who received at least 1 dose of study intervention. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 20 mg
Number analyzed (Participants) | 14
Participants
  Day 1: Taste Score: 1 | 1
  Day 1: Taste Score: 2 | 0
  Day 1: Taste Score: 3 | 3
  Day 1: Taste Score: 4 | 3
  Day 1: Taste Score: 5 | 7
  Day 1: Mouthfeel Score: 1 | 0
  Day 1: Mouthfeel Score: 2 | 5
  Day 1: Mouthfeel Score: 3 | 3
  Day 1: Mouthfeel Score: 4 | 4
  Day 1: Mouthfeel Score: 5 | 2
  Day 1: Volume Score: 1 | 2
  Day 1: Volume Score: 2 | 5
  Day 1: Volume Score: 3 | 2
  Day 1: Volume Score: 4 | 2
  Day 1: Volume Score: 5 | 3
  Day 7: Taste Score: 1 | 0
  Day 7: Taste Score: 2 | 1
  Day 7: Taste Score: 3 | 4
  Day 7: Taste Score: 4 | 2
  Day 7: Taste Score: 5 | 7
  Day 7: Mouthfeel Score: 1 | 0
  Day 7: Mouthfeel Score: 2 | 5
  Day 7: Mouthfeel Score: 3 | 3
  Day 7: Mouthfeel Score: 4 | 5
  Day 7: Mouthfeel Score: 5 | 1
  Day 7: Volume Score: 1 | 1
  Day 7: Volume Score: 2 | 6
  Day 7: Volume Score: 3 | 2
  Day 7: Volume Score: 4 | 1
  Day 7: Volume Score: 5 | 4

ADVERSE EVENTS:
Time Frame: Day 1 up to 35 days after last dose (maximum up to Day 42)
Description: Safety set evaluated.
Groups:
- Ritlecitinib 20 mg QD: Participants received Ritlecitinib 20 mg orally QD, for 7 consecutive days. Participants were followed up to 35 days after the last dose.
Arm/Group | Ritlecitinib 20 mg QD
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 3/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ritlecitinib 20 mg QD (N=15)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT05650333/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT05650333/SAP_001.pdf